CLINICAL TRIAL: NCT05516940
Title: A Study of the Impact of Different Delivery Modes on Specific Macronutrient Components in Human Milk
Acronym: ZoomMING
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Chinese Center for Disease Control and Prevention, National Institute for Nutrition and Health (Unknown); SAS Institute (Industry); Veeva Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: 21.08.NR
Record Dates: First submitted 2022-07-25; First posted 2022-08-26 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — human milk samples have already been collected within China CDC's cross sectional multi-centric human milk study conducted in China
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Caesarean-section: 125 subjects will be selected who have delivered infants by Caesarean-section.
- Normal delivery: 125 subjects will be selected who have delivered infants by vaginal/normal deliveries

INTERVENTIONS:
Other:

SUMMARY:
The aim of the study is to evaluate the impact of different delivery modes on specific macronutrient components in human milk.

DETAILED DESCRIPTION:
The main objective of the study is to explore the differences in human milk composition from mothers delivering by Caesarean-section and normal vaginal deliveries. To further associate the differences found in human milk composition to infant outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Human milk to be selected from the mothers who have delivered at full term (>37 weeks of gestation).
2. 125 subjects will be selected who have delivered infants by Caesarean-section.
3. 125 subjects will be selected who have delivered infants by vaginal/normal deliveries.
4. Subjects will be selected based on sample availability.
5. Based on sample availability to balance by stage of lactation, geographical locations within China.
6. Subjects of Han ethnicity.
7. The collection of existing biological material and/or health-related personal data have been consented in the frame of the approved original study scope. We will propose to the participants to consent to this specific research.

Exclusion Criteria:

1) Incomplete information either for the subject or the sample collected.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population of interest is mothers that have delivered at full term (>37 weeks of gestation) who have already provided human milk samples collected within China CDC's cross sectional multi-centric human milk study conducted in China.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Differences in HMO from mothers' milk who delivered by Caesarean-section and normal vaginal deliveries. | baseline (no primary mothers' milk collection, but from existing human milk samples)
  HMO will be analyzed by HPLC-FLD

SECONDARY OUTCOMES:
Differences in human milk fat from mothers who delivered by Caesarean-section and normal vaginal deliveries. | baseline (no primary collection, but from existing human milk samples)
  Fatty acid will be analyzed by GC-FID
Differences in human milk proteins from mothers who delivered by Caesarean-section and normal vaginal deliveries. | baseline (no primary collection, but from existing human milk samples)
  Proteins will be analyzed by Ultra-high phase liquid chromatography
Differences in human milk gangliosides from mothers who delivered by Caesarean-section and normal vaginal deliveries. | baseline (no primary collection, but from existing human milk samples)
  gangliosides will be analyzed by GC-MS
Association of the differences in human milk composition with subject-reported outcomes | baseline (no primary collection, but from the existing questionnaires)
  The subject-reported outcomes were existing information in the questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Center for Disease Control and Prevention, National Institute for Nutrition and Health, Beijing, China

IPD SHARING:
Plan to Share IPD: No